CLINICAL TRIAL: NCT04881435
Title: The Effect of Inhaled Hydrogen on the Prognosis of Idiopathic Sudden Sensorineural Hearing Loss
Brief Title: Hydrogen-oxygen Gas Mixture Inhalation in Patients With Sudden Sensorineural Hearing Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202000554A3
Record Dates: First submitted 2021-05-03; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrogen gas inhalation therapy accompanied with standard steroid treatment (Experimental)
  Interventions: Device: Hydrogen gas therapy
- Standard steroid treatment (Active Comparator)
  Interventions: Device: Hydrogen gas therapy

INTERVENTIONS:
Device: Hydrogen gas therapy — Hydrogen gas therapy three times one day for 5 days

SUMMARY:
Idiopathic sudden sensorineural hearing loss (ISSHL) is defined according to American Academy of Otolaryngology as a hearing loss of at least 30 decibel over 3 contiguous test frequencies occurring within a 72h period. It affects 5 to 20 people per 100,000 annually and is characterized by sudden-onset, generally unilateral, sensorineural hearing loss. Its cause is idiopathic in most of the patients; however, vascular disorders have been proposed as the final common pathway. Recent studies have reported that the impaired microvascular perfusion occurring during an ischemic event may be related to oxidative stress which may be synergistically responsible for endothelial damage, especially in terminal microvascular systems.

Hydrogen, which serves as a free radical scavenger and can reduce the strong oxidants, is found as a therapeutic gas in cochlea in recent studies. Both antioxidant and anti-inflammatory effects have been seen with hydrogen administration in animal models. Since cisplatinum toxicity and acoustic trauma both involve oxidative stress to the cochlea, hydrogen may prove useful in these conditions. The efficacy and safety of hydrogen inhalation are also proved in clinical studies.

Given the theories mentioned above, the purpose of our study is to use inhaled hydrogen as an adjuvant therapy for treating idiopathic sudden sensorineural hearing loss. The systemic inflammation status and oxidative stress will be monitored. Both subjective and objective efficacy after treatment will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the criteria of definition of sudden sensorineural hearing loss: hearing loss of 30 dB or more over at least three contiguous frequencies, over a period of 72 hours or less.
2. The event attacked within 14 days. -

Exclusion Criteria:

1. pregnancy or other vulnerable groups
2. specific etiologies of sudden sensorineural hearing loss
3. Diabetes mellitus patients -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-17 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
hearing recovery | 1.before treatment 2. after treatment immediately 3.one month later after treatment
  The level of hearing recovery between the two groups

SECONDARY OUTCOMES:
the change of systemic inflammatory status and oxidative stress | 1.before treatment 2. after treatment immediately 3.one month later after treatment
  Use some indicators of systemic inflammatory status and oxidative stress to measure the changes between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Nung Wu, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
no plan to sharing currently

REFERENCES:
- [Background] Quaranta N, De Ceglie V, D'Elia A. Endothelial Dysfunction in Idiopathic Sudden Sensorineural Hearing Loss: A Review. Audiol Res. 2016 Jul 27;6(1):151. doi: 10.4081/audiores.2016.151. eCollection 2016 Apr 20. PMID 27588164
- [Background] Gode S, Turhal G, Kaya I, Mavili HI, Kirazli T. Evaluation of Procalcitonin and hs-CRP Levels in Sudden Sensorineural Hearing Loss. J Int Adv Otol. 2018 Apr;14(1):44-47. doi: 10.5152/iao.2017.2780. Epub 2017 Jun 21. PMID 28639554
- [Background] Capaccio P, Pignataro L, Gaini LM, Sigismund PE, Novembrino C, De Giuseppe R, Uva V, Tripodi A, Bamonti F. Unbalanced oxidative status in idiopathic sudden sensorineural hearing loss. Eur Arch Otorhinolaryngol. 2012 Feb;269(2):449-53. doi: 10.1007/s00405-011-1671-2. Epub 2011 Jun 26. PMID 21706323
- [Result] Joachims HZ, Segal J, Golz A, Netzer A, Goldenberg D. Antioxidants in treatment of idiopathic sudden hearing loss. Otol Neurotol. 2003 Jul;24(4):572-5. doi: 10.1097/00129492-200307000-00007. PMID 12851547